CLINICAL TRIAL: NCT02232269
Title: Phase 1 Study of the Hemodynamic and Pharmacokinetic Interactions Between Coffee and Felodipine
Brief Title: Coffee Interaction With the Antihypertensive Drug Felodipine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, David Bailey, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R-11-655; NA-7122 (Other Grant/Funding Number: Heart & Stroke Foundation of Ontario)
Record Dates: First submitted 2014-08-28; First posted 2014-09-05 (Estimated); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Food-Drug Interactions
Keywords: Coffee; Grapefruit Juice; Felodipine; Calcium Channel Blocker; Hemodynamics; CYP3A4
MeSH Terms: interventions — Water; Felodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Water plus Felodipine (Placebo Comparator): Felodipine extended-release tablet ,10 mg, single dose, 8 hours
  Interventions: Other: Water; Drug: Felodipine
- Black Coffee (Active Comparator): Black Coffee, 300 ml, 0 and 1 hour
  Interventions: Other: Black Coffee
- Black Coffee plus Felodipine (Experimental): Black Coffee, 300 ml, 0 and 1 hour
  Felodipine extended-release tablet ,10 mg, single dose, 8 hours
  Interventions: Other: Black Coffee; Drug: Felodipine
- Grapefruit Juice plus Felodipine (Active Comparator): Grapefruit Juice, 300 ml, 0 and 1 hour
  Felodipine extended-release tablet ,10 mg, single dose, 8 hours
  Interventions: Other: Grapefruit Juice; Drug: Felodipine

INTERVENTIONS:
Other: Black Coffee
  Arms: Black Coffee; Black Coffee plus Felodipine
Other: Grapefruit Juice
  Arms: Grapefruit Juice plus Felodipine
Other: Water
  Arms: Water plus Felodipine
Drug: Felodipine
  Other Names: Plendil; Renadil
  Arms: Black Coffee plus Felodipine; Grapefruit Juice plus Felodipine; Water plus Felodipine

SUMMARY:
Coffee is a globally popular beverage. More than half of the United States population spends an estimated $ 40 billion on the purchase of coffee each year. Personal consumption habits can vary. For example, the frequency of ingestion ranged from 59% for every day to 8% for less than one day per week consumption in one survey. In the case of occasional consumption, coffee can markedly elevate blood pressure in normotensive and hypertensive individuals. This pressor effect can occur with a caffeine dose of 200 - 250 mg, which can be found 2 - 3 cups of coffee. A major active constituent in coffee is caffeine, which is the most widely used pharmacological substance in the world.

Drug therapy plays a major role in the management of hypertension. However, the interaction between coffee or caffeine and blood pressure lowering drugs has been assessed in only three clinical studies that were reported more than three decades ago.

We conducted a comprehensive interaction study involving a commonly ingested amount of a particular Colombian coffee and felodipine in healthy middle-aged men and women. Peripheral (brachial) and central (aortic) hemodynamics and caffeine and felodipine pharmacokinetics were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* healthy (normal physical exam, blood clinical chemistry)
* willingly signs ethics approved informed consent form

Exclusion Criteria:

* history of cardiac, renal, hepatic or gastrointestinal disease or substance abuse
* significant illness within 2 weeks of starting study
* history of allergy to felodipine , tablet ingredients or dihydropyridines
* routinely taking prescription or OTC drugs or natural health products
* received an investigational drug withing the previous 4 weeks
* females who are pregnant or breast-feeding

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2012-02; Primary Completion 2012-06 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
The effect of felodipine on coffee-mediated increases in peripheral and central blood pressure . | Change from Baseline to 8 hours Post Dose
  Peripheral (brachial systolic and diastolic blood pressure) and central (aortic systolic blood pressure) measurements were the mean of at least 3 readings after 5 minutes of sitting at rest. The respective instruments used were BpTRU™ Vital Signs Monitor (BpTRU Medical Devices, Coquitlam BC, Canada) and SphygmoCor® CP Pulse Wave Analysis System - Research (AtCor Medical, Inc., Itasca, IL USA).

SECONDARY OUTCOMES:
The effect of coffee on the oral pharmacokinetics of felodipine. | Change from Baseline to 8 hours Post Dose
  Area Under Curve (AUC) Time Frame: predose, 1,2,3,4,5,6,7,8 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: David G Bailey, BScPhm, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Victoria Clinical Trials Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bailey DG, Dresser GK, Urquhart BL, Freeman DJ, Arnold JM. Coffee-Antihypertensive Drug Interaction: A Hemodynamic and Pharmacokinetic Study With Felodipine. Am J Hypertens. 2016 Dec 1;29(12):1386-1393. doi: 10.1093/ajh/hpw081. PMID 27481881
- [Background] Dresser GK, Urquhart BL, Proniuk J, Tieu A, Freeman DJ, Arnold JM, Bailey DG. Coffee inhibition of CYP3A4 in vitro was not translated to a grapefruit-like pharmacokinetic interaction clinically. Pharmacol Res Perspect. 2017 Oct;5(5):e00346. doi: 10.1002/prp2.346. PMID 28971609